CLINICAL TRIAL: NCT07136129
Title: Functional Exercise Performance in Children With Cerebral Palsy: Is the One-Minute Sit-to-Stand Test an Alternative to the Six-Minute Walk Test
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Collaborators: Kayseri University (Other)
Responsible Party: Principal Investigator, Betul Ergun, research asistant, Inonu University
Other Study IDs: SP-1sts6dyt
Record Dates: First submitted 2025-07-10; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy; Cerebral Palsy Spastic Hemiplegic
Keywords: cerebral palsy; One-Minute Sit-to-Stand Test; Functional Exercise Performance in Cerebral Palsy; Six-Minute Walk Test
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spastic hemiplegic type SP: Individuals between 5 and 18 years of age, diagnosed with spastic hemiplegic type CP and in level I or II according to the Gross Motor Function Classification System (GMFCS) were included.

SUMMARY:
This study investigates the validity of the 1-minute sit-to-stand test (1MSTS) as a practical and time-efficient alternative to the 6-minute walk test (6MWT) for assessing functional exercise capacity in children with spastic cerebral palsy (CP). Children aged 5 to 18 years with spastic hemiplegic CP, classified as Level I or II according to the Gross Motor Function Classification System (GMFCS), will perform both tests on the same day. Cardiopulmonary responses and fatigue will be monitored before and after each test. The study aims to determine whether the 1MSTS can be reliably used in clinical settings as a simpler assessment tool for this population.

DETAILED DESCRIPTION:
This cross-sectional study was conducted between December 2024 and July 2025 at Kayseri City Hospital with children diagnosed with spastic hemiplegic cerebral palsy, aged 5-18 years, classified as Level I or II on the Gross Motor Function Classification System (GMFCS). Children with severe cognitive impairment, additional neurological disorders, or uncontrolled health conditions were excluded.

Participants completed both the 6-minute walk test (6MWT) and the 1-minute sit-to-stand test (1MSTS) on the same day, in random order. Tests were performed twice, and a 1-hour rest was given between them. Cardiovascular and respiratory parameters (heart rate, oxygen saturation, blood pressure), dyspnea, and leg fatigue were measured before and after each test using standard tools (pulse oximeter, sphygmomanometer, Modified Borg Scale).

The 6MWT followed ATS guidelines. The 1MSTS was performed using a height-adjustable chair without armrests, and participants stood up and sat down repeatedly for one minute. The number of completed repetitions was recorded. This study followed the Declaration of Helsinki, and written informed consent was obtained from all participants and their guardians.

ELIGIBILITY:
Inclusion Criteria:

* Having spastic hemiplegic CP between 5-18
* Being level 1 and 2 according to KMFSS

Exclusion Criteria:

* Having cognitive/mental problems at a level that may prevent communication
* Having genetic and/or neurological problems in addition to CP
* Having uncontrolled heart disease
* Having any infection Removal Criteria
* The child or his/her parents wanting to leave the study
* Failure to complete the tests to be applied within the scope of the study
* Having an additional disease/surgical operation during the study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consisted of children aged between 5 and 18 years who were diagnosed with spastic hemiplegic type cerebral palsy (CP) and were being followed up at the Physical Therapy and Rehabilitation Clinic of Kayseri City Hospital between December 2024 and July 2025. These individuals were classified as Level I or II according to the Gross Motor Function Classification System (GMFCS), indicating relatively high levels of functional mobility. All participants and their legal guardians were informed about the study's purpose and procedures, and written informed consent was obtained. The study was approved and conducted in accordance with the principles of the Declaration of Helsinki.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Number of Repetitions in the 1-Minute Sit-to-Stand Test (1MSTS) | At baseline (single assessment session)
  This outcome measures the total number of full sit-to-stand movements performed in one minute by participants with spastic hemiplegic cerebral palsy. The aim is to determine whether the 1MSTS is a valid measure of functional exercise performance in this population.
Distance Walked in the 6-Minute Walk Test (6MWT) | At baseline (single assessment session)
  Measures the total distance (in meters) walked in 6 minutes by participants on a 30-meter corridor, in accordance with ATS guidelines. The 6MWT serves as the reference test to compare with the 1MSTS.

SECONDARY OUTCOMES:
Heart Rate (HR) Before and After Exercise Tests | Pre-intervention and immediately after the intervention
  Heart rate is measured using a pulse oximeter before and after both the 1MSTS and 6MWT to assess cardiovascular response to physical activity.
Oxygen Saturation (SpO2) Before and After Exercise Tests | Pre-intervention and immediately after the intervention
  Peripheral oxygen saturation is recorded before and after each exercise test to monitor oxygenation changes in response to activity.
Systolic and Diastolic Blood Pressure Before and After Exercise Tests | Pre-intervention and immediately after the intervention
  Blood pressure values are recorded before and after the tests using a standard sphygmomanometer to evaluate cardiovascular load.
Perceived Dyspnea and Leg Fatigue Using Modified Borg Scale | Pre-intervention and immediately after the intervention
  Dyspnea and lower extremity fatigue are assessed before and after each test using the Modified Borg Scale (0-10), which evaluates subjective exertion levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided